The Mauritius and Rodrigues Non-Communicable Disease (NCD) Study

NCT07048717

Informed consent from the 2021 survey



#### MHC/CT/NETH/2020 V2

11 September 2020

From: Senior Chief Executive, Ministry of Health and Wellness

To: Dr S. Kowlessur, Chief Health Promotion and Research Coordinator

#### Request for Ethical Clearance

Please refer to your correspondence regarding the abovementioned subject and be informed that your application for Ethical Clearance in respect of the project entitled "Mauritius NCD Survey 2020/2021" has been examined at the level of the Ministry.

2. This is to inform you that the Ethics Sub-Committee has given Ethical Clearance for the above project, subject to list of conditions annexed.

Dr S. Ramen for Supervising Officer



### The National Ethics Committee

### **Decision**

**Project Protocol** 

MHC/CT/NETH/2020

**Applicant** 

Dr S. KOWLESSUR

**Project Title** 

Mauritius NCD Survey 2020/2021

The National Ethics Committee Meeting held on 10 September 2020 has

#### **Awarded Ethical Clearance**

to the above project proposal.

You are also requested to:-

- (a) submit a Progress Report every month;
- (b) notify the ethical Committee of any amendment of recruitment of material or of consent form, or of information to be submitted to the research participants;
- (c) report to the Ethical Committee any serious or unexpected, unforeseen circumstances;
- (d) report to the Ethical Committee termination of the project;
- (e) provide relevant information to the Ethical Committee for ongoing review;
- (f) give a copy of the Final Summary on the Final report to the Ethical Committee;
- (g) ensure that confidentiality is expected throughout the project; and
- (h) ensure that the question on ethnic group is optional.

Dr S. Ramen for Supervising Officer



### **MAURITIUS NON-COMMUNICABLE DISEASES SURVEY 2021**

## **Consent Form**

| | Reg. No. | |
|---|---|---|
| I, Mr/Mrs/Miss Mauritius Non-Communicable Diseases Surve and Wellness in collaboration with Baker IDI Australia; University of Helsinki, Finland; UmUK; and World Health Organization. | y 2021, which is being undertaken by<br>Heart and Diabetes Institute, Austral | the Ministry of Health<br>ia; Monash University, |
| I understand that the purpose of the survey is which include diabetes and high blood pressure consent is given voluntarily. | | |
| I agree that if results of my investigations are ab and follow up. | normal, I will be referred for further in | vestigations, treatment |
| I understand that I will be asked to provide blood and urine samples and that I will undergo physical examinations to measure my height, weight, waist, hip and neck circumferences, blood pressure, handgrip strength and pulse wave. I have been told that I will be asked some general questions about my health, lifestyle, physical activity, diet, sleep and my knowledge of good health. I have also been told that, if required, an Electrocardiogram Test, Pulse Wave Velocity Test and/or Retinal photography will be performed on me. | | |
| I have been informed that blood samples colle<br>informed that all data reporting will be done and | | |
| Name of Participant | Signature | Date |
| | | /2021 |
| Name of Witness | Signature of Witness | Date |
| | | /2021 |



### MINISTRY OF HEALTH & WELLNESS

# Mauritius Non Communicable Diseases Survey 2021

### **CERTIFICATE OF ATTENDANCE**

| | Date: |
|------------------------------------------|--------------------------------|
| Dear Sir/Madam | |
| This is to certify that Mr. /Mrs/Miss | |
| participated in the Mauritius Non Commun | icable Diseases Survey 2021 on |
| from | to hrs. |
| Your assistance in allowing him / her to | attend this survey is greatly |
| appreciated. | E HEALTH AGO. |
| With many thanks | MADRITUS (S) |
| | Copy 1-1 Observation |

**Dr. B. Ori**Director Health Services
For Ag. Senior Chief Executive